CLINICAL TRIAL: NCT01494532
Title: A Fixed Dose, Dose-response Study of Ropinirole Prolonged Release (PR) as Adjunctive Treatment to L-dopa in Patients With Advanced Parkinson's Disease
Brief Title: A Fixed Dose Study of Ropinirole Prolonged Release as Adjunctive Treatment in Patients With Advanced Parkinson's Disease
Acronym: TANDEM-569
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111569
Record Dates: First submitted 2011-12-01; First posted 2011-12-19 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ropinirole (Experimental): active treatment 4, 8, 12, 16, or 24mg/day
  Interventions: Drug: ropinirole/L-dopa
- placebo (Placebo Comparator): placebo comparator 4, 8, 12, 16, or 24mg/day
  Interventions: Drug: placebo/L-dopa

INTERVENTIONS:
Drug: ropinirole/L-dopa — Ropinirole as adjunctive therapy with L-dopa
  Arms: ropinirole
Drug: placebo/L-dopa — Placebo as adjunctive therapy with L-dopa
  Arms: placebo

SUMMARY:
This is a double blind, fixed dose, parallel group study to characterize the dose response of ropinirole PR as adjunctive therapy to L-dopa in patients with late stage Parkinson's disease. The primary endpoint of this study, mean change from baseline in total awake time spent "off' is the same endpoint as used in the ropinirole PR pivotal study for advanced Parkinson's disease patients. This study includes a wide range of ropinirole doses (4-24mg) with the 8mg, 12mg, and 16mg per day doses powered to detect a 1.7 hour difference in total awake time spent "off" compared with placebo. The dose of Ldopa will remain stable through the study, unless the subject experiences tolerability issues that require an L-dopa dose reduction. Up to three L-dopa dose reductions are allowed, making a total reduction of up to approximately 30%. Keeping the L-dopa dose constant where possible is important to avoid confounding the efficacy data. Clinical review of the primary and secondary endpoints will be performed in order to establish the lowest maximally effective therapeutic dose.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease (according to modified Hoehn & Yahr criteria Stages II-IV) and demonstrating lack of control with L-dopa therapy (e.g.

end of dose akinesia, simple on/off fluctuations).

* Subjects receiving a stable dose of L-dopa for at least 4 weeks prior to screening.
* A minimum of 3 hours awake "off-time" for each diary day recorded during the baseline period.
* Men or non-pregnant/non-breast-feeding women of at least 30 years of age at screening. Women of child-bearing potential must be practicing a clinically accepted method of contraception during the study and for at least one month prior to randomization and one month following completion of the study. Acceptable contraceptive methods include abstinence, oral contraception, injectable progestogen, implants of levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, surgical sterilisation, male partner sterilization, intrauterine device [IUD], or double barrier method: condom or occlusive cap (diaphragm or cervical/vault caps) plus spermicidal agent (foam/gel/film/cream/suppository.
* Provide written informed consent for this study.
* Be willing and able to comply with study procedures, including diary card completion and follow-up clinic visits.

Exclusion Criteria:

* Late stage advanced subjects demonstrating incapacitating peak dose or diphasic dyskinesia on their stable dose of L-dopa
* Consumption of any dopamine agonist, including ropinirole, within four weeks of randomization in the study.
* Subjects with severe, clinically significant condition(s) other than Parkinson's disease which, in the opinion of the investigator, would render the subject unsuitable for the study (e.g., psychiatric, haematological, renal, hepatic, endocrinology, neurological [other than Parkinson's disease], cardiovascular, or active malignancy [other than basal cell carcinoma]).
* Subjects with crippling degenerative arthritis or other physical or mental conditions which would preclude accurate assessment of efficacy or safety.
* Subjects with prior or current major psychosis (e.g., schizophrenia or psychotic depression) e.g. scoring 3 or 4 on UPDRS item 2 [thought disorder] or item 3 [depression].
* Subjects with severe clinical dementia e.g. scoring 3 or 4 on UPDRS item 1 [mentation].
* Subjects with severe dizziness or fainting due to postural hypotension on standing.
* Subjects with a personal history of melanoma.
* Subjects with clinically significant abnormalities in laboratory or ECG tests at Screening. If findings are outside the normal range and the subject is included, it must be documented by the investigator that the findings are not of clinical significance.
* Subjects who are diagnosed with an impulse control disorder. The modified MIDI will be conducted at screening. Subjects who score positive for this screen must be referred to a specialist for diagnostic evaluation.
* Subjects who have an active suicidal plan/intent or have had active suicidal thoughts in the past 6 months. Subjects who have a history of suicide attempt in the last 2 years or more than 1 lifetime suicide attempt.
* Current alcohol or drug dependence.
* Definite or suspected personal or family history of clinically significant adverse reactions or hypersensitivity to ropinirole (or to drugs with a similar chemical structure) that would preclude long-term dosing with ropinirole.
* Withdrawal, introduction, or change in dose of hormone replacement therapy and/or any drug known to substantially inhibit CYP1A2 (e.g. ciprofloxacine, fluvoxamine, cimetidine, ethinyloestradiol) or induce CYP1A2 (e.g. tobacco, omeprazole) within 7 days prior to enrolment (randomization). Subjects already on chronic therapy with any of these agents may be enrolled but doses must have remained stable from 7 days prior to enrolment (randomization) through the end of the treatment period.
* Women who are pregnant or breast-feeding.
* Use of an investigational drug from 30 days or 5 half-lives (whichever is longer) prior to enrolment (randomization) through to the end of the treatment period. 15. Women who are pregnant or breast-feeding. 16. Use of an investigational drug from 30 days or 5 half-lives (whichever is longer) prior to enrolment (randomization) through to the end of the treatment period.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2012-04-02 (Actual); Primary Completion 2014-11-18 (Actual); Study Completion 2014-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (41):
- United States (9):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Pasadena, California
  - GSK Investigational Site, Reseda, California
  - GSK Investigational Site, Ventura, California
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Forest Hills, New York
  - GSK Investigational Site, Richmond, Virginia
- Argentina (5):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, San Martín, Buenos Aires
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Caba
- Chile (3):
  - GSK Investigational Site, Valdivia, Los Lagos Region
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago
- GSK Investigational Site, Tallinn, Estonia
- Russia (13):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Kursk
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Saratov
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- Slovakia (4):
  - GSK Investigational Site, Banská Bystrica
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Dubnica nad Váhom
  - GSK Investigational Site, Trnava
- South Korea (6):
  - GSK Investigational Site, Anyang-si
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Seongnam-si Gyeonggi-do
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Sungnam

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 111569 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111569 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111569 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111569 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 111569 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111569 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants(par) were diagnosed with advanced stage idiopathic Parkinson's Disease (PD), demonstrated lack of control with Levo(L)-dopa therapy, and on a stable dose of L-dopa for a minimum of 4 weeks prior to screening. Par were randomized into one of six treatment arms to receive placebo or ropinirole prolonged release(PR) tablets.
Pre-assignment Details: After screening, par underwent a 13 Week up-titration period until reaching their target dose then continued on their target dose during a 4 Week Maintenance Period up to Week 17. All par underwent a 1 Week down-titration period and then a follow-up visit 2 Weeks after receiving the last dose of study medication.
Groups:
- Treatment Group A: Placebo: Participants (par.) were administered a matching prolonged release (PR) placebo tablet once daily (OD) for up to 17 Weeks followed by down titration with placebo over 1 week. Par. completed a follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group B: 4 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 milligrams per day (mg/day), OD for one week. Par. were up-titrated to 4 mg/day at Week 2 and continued this dose up to study Week 17. Par. reaching their target dose and completing the Maintenance Period or withdrawing prematurely were switched to placebo for down-titration for 1 Week before completing a follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group C: 8 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 mg/day, OD for one week. Par. were up-titrated to 4 mg/day at Week 2, 6 mg/day at Week 3, and 8 mg/day at Week 4. Par. continued this dose up to study Week 17. Par. reaching their target dose and completing the Maintenance Period or withdrawing prematurely were switched to ropinirole PR 6.0 mg/day for 4 days then 4.0 mg/day for 3 days for down-titration before completing a follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group D: 12 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 mg/day, OD for one week. Par. were up-titrated to 4 mg/day at Week 2, 6 mg/day at Week 3, 8 mg/day at Week 4 and 12 mg/day at Week 6. Par. continued this dose up to study Week 17. Par. reaching their target dose and completing the Maintenance Period or withdrawing prematurely were switched to ropinirole PR 8.0 mg/day for 4 days then 4.0 mg/day for 3 days for down-titration before completing a follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group E: 16 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 mg/day, OD for one week. Par. were up-titrated to 4 mg/day at Week 2, 6 mg/day at Week 3, 8 mg/day at Week 4, 12 mg/day at Week 6 and 16 mg/day at Week 8. Par. continued this dose up to study Week 17. Par. reaching their target dose and completing the Maintenance Period or withdrawing prematurely were switched to ropinirole PR 12.0 mg/day for 4 days then 6.0 mg/day for 3 days for down-titration before completing a follow-up visit 2 weeks after receiving the last dose of study medication.
- Treatment Group F: 24 mg/Day: Par. were administered a ropinirole PR tablet totalling 2 mg/day, OD for one week. Par. were up-titrated to 4 mg/day at Week 2, 6 mg/day at Week 3, 8 mg/day at Week 4, 12 mg/day at Week 6, 16 mg/day at Week 8, 20 mg/day at Week 10, and 24 mg/day at Week 12. Par. continued this dose up to study Week 17. Par. reaching their target dose and completing the maintenance or withdrawing prematurely were switched to ropinirole PR 16.0 mg/day for 4 days then 8.0 mg/day for 3 days for down-titration before completing a follow-up visit 2 weeks after receiving the last dose of study medication.
Period: Overall Study
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Started | 75 | 25 | 76 | 75 | 76 | 25
Completed | 65 | 21 | 59 | 60 | 64 | 25
Not Completed | 10 | 4 | 17 | 15 | 12 | 0
Not completed — Adverse Event | 4 | 1 | 8 | 6 | 5 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol deviation | 2 | 1 | 3 | 2 | 3 | 0
Not completed — Protocol-defined stopping criteria | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 4 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Group A: Placebo: Participants (par.) were administered a matching prolonged release (PR) placebo tablet once daily (OD) for up to 17 Weeks. Par. completed a follow-up visit 2 weeks after receiving the last dose of study medication.
- Total: Total of all reporting groups
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day | Total
Number analyzed (Participants) | 75 | 25 | 76 | 75 | 76 | 25 | 352
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.7 (9.98) | 66.5 (7.45) | 65.6 (9.19) | 65.2 (9.62) | 63.7 (9.13) | 66.9 (7.94) | 64.8 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 12 | 33 | 33 | 38 | 10 | 168
  Male | 33 | 13 | 43 | 42 | 38 | 15 | 184
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 2 | 0 | 0 | 0 | 0 | 0 | 2
  American Indian or Alaskan Native | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian - East Asian Heritage | 3 | 3 | 3 | 4 | 6 | 1 | 20
  Asian - Japanese Heritage | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian - South East Asian Heritage | 0 | 1 | 0 | 1 | 1 | 0 | 3
  White - White/Caucasian/European Heritage | 70 | 21 | 73 | 68 | 69 | 24 | 325

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (BL) in Total Awake Time Spent "Off" at Week 4 of Maintenance Period
Description: "Off" time is defined as the state in which the participants(par) symptoms include lack of mobility(bradykinesia) with or without additional features such as tremor or rigidity. Par were asked to record awake time "off ", awake time "on", troublesome dyskinesias(TD) during awake time "on", or time asleep for 30 minute intervals in 24 hr diary cards for 2 days preceding visits. Total number of awake hrs spent "off" per 24-hr period was the average of the 2 diary cards of the sum of awake hours spent "off" in each 24-hr diary card. BL is the last non-missing assessment measured on or before the first dose, change from BL was calculated by subtracting the BL values from the MP Week 4 values. Mixed Model Repeated Measures (MMRM) model used BL total awake time 'Off', treatment, visit and treatment by visit
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: The Intent to Treat(ITT) Population included all randomized par who received at least one dose of study medication, had a BL efficacy assessment for the outcome, and at least one respective Post-BL efficacy assessment. Participants with a non-missing efficacy observation at Baseline and during the maintenance period were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Groups:
- Treatment Group A: Placebo: Participants (par.) were administered matching prolonged release (PR) placebo tablet once daily (OD) for up to 17 Weeks followed by down titration with placebo over 1 week. Par. completed a follow-up visit 2 weeks after receiving the last dose of study medication.
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Hours | -1.91 [-2.46 to -1.35] | -2.04 [-3.02 to -1.06] | -2.92 [-3.50 to -2.34] | -2.34 [-2.91 to -1.76] | -2.80 [-3.36 to -2.24] | -2.37 [-3.26 to -1.47]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; 4mg/day vs Placebo; Test type: Superiority or Other; p = 0.814, Mixed Models Analysis — P-values were estimated from Mixed Model Repeated Measures (MMRM)
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; 8 mg/day vs Placebo; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — P-values were estimated from Mixed Model Repeated Measures (MMRM)
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; 12 mg/day vs Placebo; Test type: Superiority or Other; p = 0.287, Mixed Models Analysis — P-values were estimated from Mixed Model Repeated Measures (MMRM)
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; 16 mg/day vs Placebo; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis — P-values were estimated from Mixed Model Repeated Measures (MMRM)
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; 24 mg/day vs Placebo; Test type: Superiority or Other; p = 0.390, Mixed Models Analysis — P-values were estimated from Mixed Model Repeated Measures (MMRM)
Statistical Analysis 6: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; 4mg/day vs Placebo; Test type: Superiority or Other; p = 0.844, ANCOVA — P-values are from a nonparametric rank ANCOVA
Statistical Analysis 7: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; 8 mg/day vs Placebo; Test type: Superiority or Other; p = 0.030, ANCOVA — P-values are from a nonparametric rank ANCOVA
Statistical Analysis 8: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; 12 mg/day vs Placebo; Test type: Superiority or Other; p = 0.437, ANCOVA — P-values are from a nonparametric rank ANCOVA
Statistical Analysis 9: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; 16 mg/day vs Placebo; Test type: Superiority or Other; p = 0.034, ANCOVA — P-values are from a nonparametric rank ANCOVA
Statistical Analysis 10: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; 24 mg/day vs Placebo; Test type: Superiority or Other; p = 0.808, ANCOVA — P-values are from a nonparametric rank ANCOVA

2. Secondary Outcome: Responder Rate Defined as the Percentage of Participants With a 20% Reduction in Baseline (BL) "Off" Time at Week-4 of Maintenance Period
Description: The responder rate was defined as the percentage of par with greater than or equal to (>=) 20 percent (%) reduction in their individual BL "off" time at Week 4 of the Maintenance Period. The "off" time is defined as the state in which the participants' symptoms include lack of mobility (bradykinesia) with or without additional features such as tremor or rigidity. BL is defined as the last non-missing assessment measured on or before the first dose date. Responder Rate (Least Squares [LS] means on inverse linked scale), odds ratio with 95% CI and p-value comparing against placebo were estimated by Generalized Estimating Equations (GEE) model. Baseline total awake time 'Off', treatment, visit and treatment*visit are included in the model.
Time Frame: Week 4 of the Maintenance Period (Study Week 17)
Population: ITT Population. Participants with a non-missing efficacy observation at Baseline and during the maintenance period were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
percentage of participants | 65.4 [52.4 to 76.4] | 68.0 [46.6 to 83.8] | 75.4 [63.0 to 84.6] | 64.3 [50.8 to 75.8] | 77.9 [66.0 to 86.5] | 72.0 [51.1 to 86.4]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.826, Generalized Estimating Equations model; Odds Ratio (OR) = 1.123, 95% CI 2-sided [0.398 to 3.166]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.233, Generalized Estimating Equations model; Odds Ratio (OR) = 1.622, 95% CI 2-sided [0.732 to 3.593]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.902, Generalized Estimating Equations model; Odds Ratio (OR) = 0.953, 95% CI 2-sided [0.439 to 2.065]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.127, Generalized Estimating Equations model; Odds Ratio (OR) = 1.866, 95% CI 2-sided [0.837 to 4.158]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.564, Generalized Estimating Equations model; Odds Ratio (OR) = 1.362, 95% CI 2-sided [0.477 to 3.888]

3. Secondary Outcome: Percentage of Participants With a >=1 Hour Reduction in Baseline "Off" Time at Week 4 of the Maintenance Period
Description: The "off" time is defined as the state in which the participants' symptoms include lack of mobility (bradykinesia) with or without additional features such as tremor or rigidity. BL is defined as the last non-missing assessment measured on or before the first dose date. The percent change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. Percentage of participants meeting the criterion (LS mean on inverse linked scale), odds ratio with 95% CI and p-value comparing against placebo were estimated by Generalized Estimating Equations (GEE) model. Baseline 'off-time', treatment, visit and treatment*visit are included in the model.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
percentage of participants | 72.1 [59.5 to 82.0] | 70.1 [48.6 to 85.4] | 80.6 [68.7 to 88.7] | 73.5 [59.6 to 83.9] | 83.2 [72.1 to 90.5] | 81.4 [62.3 to 92.0]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.861, Generalized Estimating Equations model; Odds Ratio (OR) = 0.908, 95% CI 2-sided [0.310 to 2.659]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.277, Generalized Estimating Equations model; Odds Ratio (OR) = 1.608, 95% CI 2-sided [0.684 to 3.782]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.869, Generalized Estimating Equations model; Odds Ratio (OR) = 1.074, 95% CI 2-sided [0.461 to 2.500]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.140, Generalized Estimating Equations model; Odds Ratio (OR) = 1.916, 95% CI 2-sided [0.808 to 4.545]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.362, Generalized Estimating Equations model; Odds Ratio (OR) = 1.689, 95% CI 2-sided [0.547 to 5.218]

4. Secondary Outcome: Percentage of Participants With a >=2 Hours Reduction in Baseline "Off" Time at Week 4 of the Maintenance Period
Description: as for outcome 3
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
percentage of participants | 53.7 [39.8 to 67.1] | 45.6 [26.8 to 65.8] | 68.2 [54.8 to 79.2] | 53.6 [39.3 to 67.3] | 63.2 [49.6 to 75.0] | 51.3 [30.1 to 72.0]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.525, Generalized Estimating Equations model; Odds Ratio (OR) = 0.723, 95% CI 2-sided [0.266 to 1.965]
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.130, Generalized Estimating Equations model; Odds Ratio (OR) = 1.851, 95% CI 2-sided [0.834 to 4.109]
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.992, Generalized Estimating Equations model; Odds Ratio (OR) = 0.996, 95% CI 2-sided [0.444 to 2.232]
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.329, Generalized Estimating Equations model; Odds Ratio (OR) = 1.480, 95% CI 2-sided [0.674 to 3.248]
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.856, Generalized Estimating Equations model; Odds Ratio (OR) = 0.907, 95% CI 2-sided [0.315 to 2.610]

5. Secondary Outcome: Responder Rate According to the Clinical Global Impression-global Improvement (CGI-I) Scale at Week 4 of the Maintenance Period
Description: The CGI-I scale allows the investigator to rate the participant's total improvement since the beginning of treatment (Baseline). Baseline is defined as the last non-missing assessment measured on or before the first dose date. The scale is rated from 1-7 where 1 = "very much improved", 2 = "much improved", 3 = "minimally improved", 4 = "no change", 5 = "minimally worse, 6 = "much worse", and 7 = "very much worse". The responder rate is defined as the percentage of participants with a score of 1 or 2. The Generalized Estimating Equations (GEE) model was used to determine CGI responder rate with treatment, visit, and treatment by visit interaction included in the model. Only scheduled visits were included.
Time Frame: Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of participants | 35 | 28 | 39 | 42 | 46 | 56

6. Secondary Outcome: Change From Baseline in Absolute Awake Time Spent "on" Without Troublesome Dyskinesia (TD) at Week 4 of the Maintenance Period
Description: Dyskinesias are involuntary twisting, turning movements caused by medication during "on" time in Parkinson's Disease (PD). TD is defined as those movements that interfere with function and cause meaningful discomfort. Par were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit. The total number of awake hours spent "on" without TD per 24-hour period was the average across the 2 diary cards of the sum of awake hours spent "on" without TD in each 24 hour diary card. The change from BL was calculated by subtracting the BL values from the MP Week 4 values. LS means, 95% CIs and P-values were estimated from Mixed Model Repeated Measures (MMRM). Par with a non-missing efficacy observation at BL and during the MP were analyzed.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Hours | 1.76 [1.15 to 2.36] | 1.21 [0.15 to 2.27] | 2.69 [2.06 to 3.31] | 2.16 [1.54 to 2.78] | 2.49 [1.89 to 3.10] | 2.24 [1.27 to 3.21]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.376, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.362, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.089, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.403, Mixed Models Analysis — Mixed Model Repeated Measures

7. Secondary Outcome: Change From Baseline in Absolute Awake Time Spent "on" at Week 4 of the Maintenance Period
Description: Par were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total number of awake hours spent "on" per 24-hour period was the average across the 2 diary cards of the sum of the awake hours spent "on" in each 24 hour diary card. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Hours | 1.70 [1.10 to 2.30] | 1.20 [0.14 to 2.25] | 2.69 [2.06 to 3.31] | 2.23 [1.61 to 2.85] | 2.62 [2.02 to 3.23] | 2.34 [1.38 to 3.31]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.419, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.230, Mixed Models Analysis
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.266, Mixed Models Analysis — Mixed Model Repeated Measures

8. Secondary Outcome: Change From Baseline for Total Sleep Time During the Night Time Hours of Sleep at Week 4 of the Maintenance Period
Description: Par. were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total sleep hours during the night time hours of sleep was the average across the 2 diary cards of the sum of time (hours) asleep during night time in each 24-hour diary card. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Hours | 0.22 [-0.13 to 0.56] | 0.86 [0.25 to 1.46] | 0.22 [-0.14 to 0.58] | 0.15 [-0.21 to 0.51] | 0.14 [-0.21 to 0.49] | 0.04 [-0.51 to 0.60]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.073, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.996, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.791, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.747, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.600, Mixed Models Analysis — Mixed Model Repeated Measures

9. Secondary Outcome: Percent Change From Baseline in Awake Time Spent "Off" at Week 4 of the Maintenance Period
Description: The "off" state is defined as the state in which the participants' symptoms include lack of mobility (bradykinesia), with or without additional features such as tremor or rigidity. Par. were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total number of awake hours spent "off" per 24-hour period was the average across the 2 diary cards of the sum of awake hours spent "off" in each 24-hour diary card. The percent change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values divided by BL values multiplied (×) the results with 100. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "off" time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "off" time in hours | -30.44 [-39.67 to -21.21] | -30.47 [-46.69 to -14.24] | -46.65 [-56.27 to -37.03] | -37.26 [-46.81 to -27.71] | -48.36 [-57.64 to -39.08] | -34.37 [-49.23 to -19.50]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.998, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.017, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.312, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.659, Mixed Models Analysis — Mixed Model Repeated Measures

10. Secondary Outcome: Percent Change From Baseline in Awake Time Spent "on" Without TD at Week 4 of the Maintenance Period
Description: Dyskinesias are involuntary twisting, turning movements caused by medication during "on" time in PD. TD is defined as those movements that interfere with function and cause meaningful discomfort. Par. were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total number of awake hours spent "on" without TD per 24-hour period was the average across the 2 diary cards of the sum of awake hours spent "on" without TD in each 24-hour diary card. The percent change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values divided by BL values × 100. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "on" time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "on" time in hours | 24.55 [15.05 to 34.04] | 15.20 [-1.37 to 31.78] | 35.20 [25.38 to 45.02] | 32.02 [22.20 to 41.84] | 34.45 [24.94 to 43.97] | 29.58 [14.39 to 44.76]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.337, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.126, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.283, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.148, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.581, Mixed Models Analysis — Mixed Model Repeated Measures

11. Secondary Outcome: Percent Change From Baseline in Awake Time Spent "on" at Week 4 of the Maintenance Period
Description: Par. were asked to recordawake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total number of awake hours spent "on" per 24-hour period was the average across the 2 diary cards of the sum of awake hours spent "on" in each 24-hour diary card. The percent change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values divided by BL values × 100. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "on" time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "on" time in hours | 21.31 [12.53 to 30.09] | 15.05 [-0.28 to 30.38] | 35.68 [26.60 to 44.77] | 31.28 [22.19 to 40.36] | 32.34 [23.60 to 41.08] | 32.43 [18.39 to 46.48]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.486, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.121, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.081, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.187, Mixed Models Analysis — Mixed Model Repeated Measures

12. Secondary Outcome: Percent Change From Baseline in Total Sleep Time During the Night Time Hours of Sleep, at Week 4 of the Maintenance Period
Description: Par. were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total sleep hours during the night time hours of sleep was the average across the 2 diary cards of the sum of time (hours) asleep during night time in each 24-hour diary card. BL is defined as the last non-missing assessment measured on or before the first dose date. The percent change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values divided by BL value × 100. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of total sleep time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of total sleep time in hours | 3.99 [-0.42 to 8.39] | 10.79 [3.04 to 18.54] | 4.94 [0.34 to 9.54] | 3.41 [-1.15 to 7.98] | 3.60 [-0.83 to 8.03] | 0.91 [-6.19 to 8.01]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.134, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.768, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.859, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.903, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.470, Mixed Models Analysis — Mixed Model Repeated Measures

13. Secondary Outcome: Change From Baseline in the Percent Awake Time Spent "Off" at Week 4 of the Maintenance Period
Description: The "off" state is defined as the state in which the participants' symptoms include lack of mobility(bradykinesia), with or without additional features such as tremor or rigidity. Par were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total number of awake hours spent "off" per 24-hour period was the average across the 2 diary cards of the sum of awake hours spent "off" in each 24-hour diary card. The percentage of awake time spent "off"= Awake time spent "off" divided by (Awake time spent "off" + Awake time spent "on") × 100. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the MP Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "off" time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "off" time in hours | -12.43 [-16.03 to -8.84] | -11.60 [-17.93 to -5.27] | -18.41 [-22.16 to -14.66] | -15.36 [-19.08 to -11.64] | -17.81 [-21.43 to -14.20] | -15.01 [-20.81 to -9.22]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.822, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.267, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.458, Mixed Models Analysis — Mixed Model Repeated Measures

14. Secondary Outcome: Change From Baseline in the Percent Awake Time Spent "on" Without TD at Week 4 of the Maintenance Period
Description: Dyskinesias are involuntary twisting, turning movements caused by medication during "on" time in PD. TD is defined as those movements that interfere with function and cause meaningful discomfort. Par were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hr diary cards for the 2 days preceding each visit of the study. The total number of awake hr spent "on" without TD per 24-hr period was the average across the 2 diary cards of the sum of awake hr spent "on" without TD in each 24-hr diary card. Percentage of awake time spent "on"without TD= Awake time spent "on" without TD divided by(Awake time spent "on" + Awake time spent "off") × 100. BL is defined as the last non-missing assessment measured on or before the first dose date, change from BL was calculated by subtracting BL values from MP Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "on" time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "on" time in hours | 12.89 [9.15 to 16.62] | 11.58 [5.01 to 18.15] | 18.34 [14.44 to 22.24] | 14.99 [11.12 to 18.85] | 17.05 [13.30 to 20.80] | 14.56 [8.54 to 20.59]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.734, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.048, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.443, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.123, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.641, Mixed Models Analysis — Mixed Model Repeated Measures

15. Secondary Outcome: Change From Baseline in the Percent Awake Time Spent "on" at Week 4 of the Maintenance Period
Description: Par. were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total number of awake hours spent "on" per 24-hour period was the average across the 2 diary cards of the sum of awake hours spent "on" in each 24-hour diary card. The percentage of awake time spent "on"= Awake time spent "on" divided by (Awake time spent "on" + Awake time spent "off") × 100. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "on" time in hours
Groups:
- Treatment Group A: Placebo: Participants (par.) were administered matching prolonged release (PR) placebo tablet once daily (OD) for up to 17 Weeks. Par. completed a follow-up visit 2 weeks after receiving the last dose of study medication.
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "on" time in hours | 12.43 [8.84 to 16.03] | 11.60 [5.27 to 17.93] | 18.41 [14.66 to 22.16] | 15.36 [11.64 to 19.08] | 17.81 [14.20 to 21.43] | 15.01 [9.22 to 20.81]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.822, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.267, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.458, Mixed Models Analysis — Mixed Model Repeated Measures

16. Secondary Outcome: Change From Baseline in the Percent of a 24-hour Day Spent "Off" at Week 4 of the Maintenance Period
Description: The "off" state is defined as the state in which the participants' symptoms include lack of mobility (bradykinesia), with or without additional features such as tremor or rigidity. Par were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total number of day awake hours spent "off" per 24-hour period was the average across the 2 diary cards of the sum of awake hours spent "off" in each 24-hour diary card. The percentage of 24 hour day spent "off"= awake time spent "off" divided by 24 x 100. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the MP Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "off" time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "off" time in hours | -7.94 [-10.26 to -5.62] | -8.50 [-12.57 to -4.43] | -12.17 [-14.59 to -9.76] | -9.75 [-12.14 to -7.35] | -11.65 [-13.98 to -9.32] | -9.86 [-13.59 to -6.13]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.814, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.287, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.027, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.390, Mixed Models Analysis — Mixed Model Repeated Measures

17. Secondary Outcome: Change From Baseline in the Percent of a 24- Hour Day Spent "on" Without TD at Week 4 of the Maintenance Period
Description: Dyskinesias are involuntary twisting, turning movements caused by medication during "on" time in PD. TD is defined as those movements that interfere with function and cause meaningful discomfort. Par were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hr diary cards for the 2 days preceding each visit. The total number of day awake hr spent "on" without TD per 24-hr period was the average across the 2 diary cards of the sum of awake hours spent "on" without TD in each 24-hour diary card. The percentage of 24 hr day spent "on" without TD= awake time spent "on" without TD divided by 24 × 100. BL is defined as the last non-missing assessment measured on or before the first dose date, change from BL was calculated by subtracting the BL values from the MP Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "on" time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "on" time in hours | 7.32 [4.81 to 9.83] | 5.03 [0.62 to 9.44] | 11.19 [8.57 to 13.81] | 8.99 [6.40 to 11.59] | 10.40 [7.88 to 12.91] | 9.34 [5.30 to 13.38]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.376, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.362, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.089, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.403, Mixed Models Analysis — Mixed Model Repeated Measures

18. Secondary Outcome: Change From Baseline in the Percent of a 24-hour Day Spent "on" at Week 4 of the Maintenance Period
Description: Par. were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total number of day awake hours spent "on" per 24-hour period was the average across the 2 diary cards of the sum of awake hours spent "on" in each 24-hour diary card. The percentage of a 24-hour day spent "on" = Awake time spent "on" divided by 24 × 100. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of "on" time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of "on" time in hours | 7.08 [4.57 to 9.58] | 4.99 [0.59 to 9.39] | 11.20 [8.59 to 13.81] | 9.28 [6.69 to 11.87] | 10.94 [8.42 to 13.45] | 9.76 [5.73 to 13.80]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.419, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.026, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.230, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.033, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.266, Mixed Models Analysis — Mixed Model Repeated Measures

19. Secondary Outcome: Change From Baseline in Total Sleep Time During the Night Time Hours of Sleep as a Percentage of a 24-hour Day, at Week 4 of the Maintenance Period
Description: Par were asked to record awake time "off", awake time "on", TD during awake time "on", or time asleep for all 30 minute time intervals in 24 hour diary cards for the 2 days preceding each visit of the study. The total sleep hours during the night time hours of sleep was the average across the 2 diary cards of the sum of time (hours) asleep during night time in each 24-hour diary card. The percentage of a 24-hour day spent asleep during the night time hours = Total sleep hours during the night time hours of sleep divided by 24 × 100. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of time in hours
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Percentage of time in hours | 0.91 [-0.53 to 2.35] | 3.57 [1.04 to 6.10] | 0.92 [-0.59 to 2.42] | 0.63 [-0.86 to 2.12] | 0.58 [-0.87 to 2.02] | 0.18 [-2.14 to 2.50]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.073, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.996, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.791, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.747, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.600, Mixed Models Analysis — Mixed Model Repeated Measures

20. Secondary Outcome: Change From Baseline in Unified Parkinson Disease Rating Scale (UPDRS) Motor Score With Participants in an "on" State, at Week 4 of the Maintenance Period
Description: The UPDRS is a clinician based rating scale used to measure motor impairments and disability. The UPDRS assesses six features of PD impairment. These are evaluated using a combination of data collected by interview and examination of the par.. One of the six features include the Part III-motor examination where scores can range 0 to 108 with par. in an "on" state where the maximum score indicates the worse condition. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 64 | 21 | 59 | 60 | 65 | 24
Score on scale | -4.75 [-6.78 to -2.72] | -10.38 [-13.94 to -6.82] | -8.43 [-10.54 to -6.32] | -8.34 [-10.43 to -6.24] | -8.86 [-10.88 to -6.85] | -10.06 [-13.37 to -6.75]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.014, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.016, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — Mixed Model Repeated Measures

21. Secondary Outcome: Change From Baseline in UPDRS Activities of Daily Living (ADL) Score With Participants in an "on" State, at Week 4 of the Maintenance Period
Description: The UPDRS Part II is the ADL score and can range from 0 to 52 as determined by the physician. The higher score indicates the worse condition. Test were performed when the par. is in the "on" state of PD. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 20 | 60 | 58 | 63 | 24
Score on scale | -1.32 [-2.17 to -0.47] | -3.08 [-4.61 to -1.56] | -3.06 [-3.94 to -2.18] | -2.18 [-3.07 to -1.28] | -2.63 [-3.49 to -1.77] | -3.04 [-4.43 to -1.65]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.047, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.005, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.172, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.034, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis — Mixed Model Repeated Measures

22. Secondary Outcome: Change From Baseline in UPDRS ADL Score With Participants in an "Off" State, at Week 4 of the Maintenance Period
Description: The UPDRS Part II is the ADL score and can range from 0 to 52 as determined by the physician. The higher score indicates the worse condition. Test was performed when the par is in the "off" state of PD. The "off" time is defined as the state in which the participants' symptoms include lack of mobility (bradykinesia) with or without additional features such as tremor or rigidity. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the Maintenance Period Week 4 values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 62 | 15 | 52 | 50 | 57 | 22
Score on scale | -2.94 [-4.23 to -1.65] | -4.50 [-7.12 to -1.88] | -4.72 [-6.13 to -3.31] | -4.29 [-5.74 to -2.84] | -5.76 [-7.11 to -4.41] | -4.77 [-6.94 to -2.61]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.292, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.068, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.170, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.153, Mixed Models Analysis — Mixed Model Repeated Measures

23. Secondary Outcome: Change From Baseline in UPDRS Part I at Week 4 of the Maintenance Period
Description: The UPDRS Part I scores mentation, behavior and mood as determined by a physician and par. were tested during the "on" phase of PD. This component of the UPDRS is the total score for 4 items (the items 1 to 4 include intellectual impairment, thought disorder, motivation / initiative, and depression) and may have a value ranging from 0 to 16 as determined by a physician. The higher score (16) indicates the maximum score and the worse condition. All 4 items have to be present for a total score to be calculated. If one or more items are missing, the total score for the component would also be missing. BL is defined as the last non-missing assessment measured on or before the first dose date. The change from BL was calculated by subtracting the BL values from the individual post-randomization values. LS means, 95% CIs and P-values were estimated from MMRM.
Time Frame: Baseline (BL) and Week 4 of the Maintenance Period (Study Week 17)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on scale
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 65 | 21 | 60 | 61 | 65 | 25
Score on scale | -0.24 [-0.47 to -0.01] | -0.44 [-0.84 to -0.03] | -0.33 [-0.57 to -0.09] | -0.24 [-0.48 to -0.00] | -0.47 [-0.70 to -0.24] | -0.45 [-0.82 to -0.08]
Statistical Analysis 1: Comparison: Treatment Group A: Placebo vs Treatment Group B: 4 mg/Day; Test type: Superiority or Other; p = 0.409, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 2: Comparison: Treatment Group A: Placebo vs Treatment Group C: 8 mg/Day; Test type: Superiority or Other; p = 0.598, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 3: Comparison: Treatment Group A: Placebo vs Treatment Group D: 12 mg/Day; Test type: Superiority or Other; p = 0.992, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 4: Comparison: Treatment Group A: Placebo vs Treatment Group E: 16 mg/Day; Test type: Superiority or Other; p = 0.169, Mixed Models Analysis — Mixed Model Repeated Measures
Statistical Analysis 5: Comparison: Treatment Group A: Placebo vs Treatment Group F: 24 mg/Day; Test type: Superiority or Other; p = 0.348, Mixed Models Analysis — Mixed Model Repeated Measures

24. Secondary Outcome: Percentage of Participants Withdrawn From the Study Due to Lack of Efficacy
Description: The percentage of participants who withdrew from the study due to lack of efficacy as defined by either the participant or the investigator is presented here. All participants with a non-missing efficacy observation at Baseline and at least one post-Baseline efficacy assessment at any time during the study were analyzed.
Time Frame: From start of study treatment until end of treatment (assessed up to 18 weeks)
Population: ITT Population. Participants with a non-missing efficacy observation at Baseline and at least one post-Baseline efficacy assessment at any time during the study were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Number analyzed (Participants) | 74 | 25 | 76 | 73 | 76 | 25
Percentage of participants | 0 | 0 | 0 | 0 | 3 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the initial dose of study treatment through the completion of the Follow-up Period (up to 33 Weeks)
Description: On-treatment SAEs and non-serious AEs were reported for the Safety Population, comprised all participants exposed to at least one dose of study medication.
Arm/Group | Treatment Group A: Placebo | Treatment Group B: 4 mg/Day | Treatment Group C: 8 mg/Day | Treatment Group D: 12 mg/Day | Treatment Group E: 16 mg/Day | Treatment Group F: 24 mg/Day
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/25 | 3/76 | 0/75 | 1/76 | 0/25
Other Adverse Events (participants affected / at risk) | 31/75 | 9/25 | 27/76 | 40/75 | 43/76 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group A: Placebo (N=75) | Treatment Group B: 4 mg/Day (N=25) | Treatment Group C: 8 mg/Day (N=76) | Treatment Group D: 12 mg/Day (N=75) | Treatment Group E: 16 mg/Day (N=76) | Treatment Group F: 24 mg/Day (N=25)
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hernia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Impulsive behaviour (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group A: Placebo (N=75) | Treatment Group B: 4 mg/Day (N=25) | Treatment Group C: 8 mg/Day (N=76) | Treatment Group D: 12 mg/Day (N=75) | Treatment Group E: 16 mg/Day (N=76) | Treatment Group F: 24 mg/Day (N=25)
Constipation (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 1 | 5 | 8 | 7 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0 | 2 | 2 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 4 | 0 | 1 | 3 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 2 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 3 | 6 | 4 | 1
Dyskinesia (Nervous system disorders) | 1 | 1 | 3 | 5 | 8 | 1
Headache (Nervous system disorders) | 4 | 0 | 2 | 3 | 4 | 1
Somnolence (Nervous system disorders) | 4 | 1 | 4 | 9 | 8 | 0
Sudden onset of sleep (Nervous system disorders) | 2 | 2 | 4 | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 4 | 0
Hypertension (Vascular disorders) | 1 | 2 | 1 | 1 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.